CLINICAL TRIAL: NCT01534000
Title: Cardiac-CT in the Treatment of Acute Chest Pain
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jens D Hove, MD,PHD, Chief of Cardiac CT, MD,PHD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-C-2009-053
Record Dates: First submitted 2011-12-22; First posted 2012-02-16 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Ischemic Heart Disease
Keywords: Cardiac CT; Ischemic heat disease; Stress test
MeSH Terms: conditions — Myocardial Ischemia | interventions — Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT guided group (Active Comparator): For Patients with chest pain randomised to this arm, clinical decision will be based on the results of a Cardiac computed tomographic angiography (CCTA)
  Interventions: Procedure: Cardiac computed tomographic angiography (CCTA)
- Control group (No Intervention): Patients with chest pain randomised to the control group will be evaluated using the standard functional-based strategy with either a treadmill stress-test or SPECT (single-photon emission computed tomography). A Cardiac CT will will be performed, but will be blinded for initial clinical evaluation.

INTERVENTIONS:
Procedure: Cardiac computed tomographic angiography (CCTA) — Patients will (on top of the standard clinical evaluation with a functional-based stress-test) be examined with a Cardiac CT scan. In the control group, the Cardiac CT will be blinded for clinical evaluation and only used retrospectively for research purpose.
  Other Names: Adenosin for CT myocardial perfusion
  Arms: CT guided group

SUMMARY:
Objectives The CATCH trial (CArdiac cT in the treatment of acute CHest pain) is a prospective randomized controlled trial designed to evaluate the clinical value of cardiac multidetector computed tomography (MDCT) as a first-line diagnostic strategy in patients with acute chest pain, compared to a conventional functional-based testing strategy.

Methods:

Consecutive patients admitted with acute chest pain of suspected cardiac origin, but normal electrocardiogram and biomarkers were randomized to evaluation with 320-MDCT coronary angiography (CT-guided group) or with standard bicycle exercise test and/or myocardial perfusion imaging - MPI (Control group).

After one year, patients will be followed-up, with registration of clinical endpoints such as Cardiac death, myocardial infarction, need for revascularisation, admittance for heart related problems, sustained chest pain, live quality score, use of medication.

ELIGIBILITY:
Inclusion Criteria:

* Admittance because of Chest pain
* Non- or non-diagnostic ecg-changes.
* Normal biomarkers for ischemia (Troponins)
* Chest X-ray without pathological findings associated with chest pain.

Exclusion Criteria:

* Women of childbearing age, or > 40 years and using approved contraception.
* Claustrophobia
* Patients with geographical residence, that complicates follow-up
* Patients with mental or physical conditions that impede follow-up
* Increase in Troponins
* New diagnostic ECG changes with ST-segment elevation or depression greater than 1mm or T-yew inversion> 4 mm in> 2 anatomically connected derivations.
* Allergy to iodinated contrast agents
* Serum creatinine greater than 130 mg/l
* Abnormal chest x-ray or blood tests hospitalization as assessed as the main cause of the patient's pain problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
combined endpoint of: Cardiac death, myocardial infarction, unstabile angina, revascularisation, readmissions for chest pain | 1 year follow-up

SECONDARY OUTCOMES:
Cardiac death | 1 year follow-up
myocardial infarction | 1 year follow-up
readmissions for chest pain | 1 year follow-up
Revascularisation | 1 year follow-up
unstabile angina | 1-year follow-up
continued chest pain | 1 year follow-up
Quality of life (SF-36) | 1-year follow-up
medication | 1-year follow-up
non-cardiac findings on CT | 1-year follow-up
downstream testing | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jesper J Linde, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Linde JJ, Hove JD, Sorgaard M, Kelbaek H, Jensen GB, Kuhl JT, Hindso L, Kober L, Nielsen WB, Kofoed KF. Long-Term Clinical Impact of Coronary CT Angiography in Patients With Recent Acute-Onset Chest Pain: The Randomized Controlled CATCH Trial. JACC Cardiovasc Imaging. 2015 Dec;8(12):1404-1413. doi: 10.1016/j.jcmg.2015.07.015. Epub 2015 Nov 11. PMID 26577263